CLINICAL TRIAL: NCT01991613
Title: Early Liquid Protein Supplementation of Human Milk in Extremely Low Birth Weight Infants
Brief Title: Early Protein Supplementation of Human Milk in Extremely Low Birth Weight Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Andrea Weintraub, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-1422
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Growth in Premature Infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- liquid protein supplement (Experimental): Study subjects will receive standard of care nutrition with the addition of a liquid protein supplement when the baby is able to tolerate an enteral feeding volume of 40mL/kg/day.
  Interventions: Dietary Supplement: liquid protein supplement
- Control group (No Intervention): Study subjects will receive standard of care nutrition

INTERVENTIONS:
Dietary Supplement: liquid protein supplement — The liquid protein supplement is already in use. The purpose of this study is to determine whether using the supplement earlier will lead to improved growth.
  Other Names: Abbott liquid protein supplement
  Arms: liquid protein supplement

SUMMARY:
We hypothesize that premature infants who receive their mothers' expressed breast milk supplemented with liquid protein early in their hospitalization will have a growth velocity in the first 28 days of life that is 20% greater than the growth velocity of premature infants that do not receive protein fortification.

ELIGIBILITY:
Inclusion Criteria:

* inborn at Mount Sinai Medical Center
* gestational age between 26 0/7 weeks and 32 6/7 weeks gestation
* plan by family for their infant to receive human milk feeds

Exclusion Criteria:

* outborn infants
* gestational age < 26 0/7 weeks or > 33 0/7 weeks
* major congenital anomalies including cardiac disease, inborn errors of metabolism etc.
* sepsis and/or other serious clinical complication precluding initiation of enteral feeds
* plan by family for their infant to receive primarily preterm infant formula.

Ages: 26 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Growth velocity | up to 28 days
  Growth velocity over the first 28 days of life - Daily weight measurements for the first 28 days of life

SECONDARY OUTCOMES:
weight | average 11 weeks
  Extrauterine growth from birth until discharge from the NICU - Weekly weight measurements until discharge from the NICU
Length | average 11 weeks
  Extrauterine growth from birth until discharge from the NICU - Weekly length measurements until discharge from the NICU
head circumference | average 11 weeks
  Extrauterine growth from birth until discharge from the NICU - Weekly head circumference measurements until discharge from the NICU

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Weintraub, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States